CLINICAL TRIAL: NCT01171547
Title: Daptomycin Pharmacokinetics in Critically Ill Patients Undergoing Continuous Veno-venous Hemodiafiltration, a Dose Find Study
Brief Title: Daptomycin Pharmacokinetics in Continuous Veno-venous Hemodiafiltration
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Prof. Marco Maggiorini, MD, Medical Intensive Care Unit
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: EK-1632
Record Dates: First submitted 2010-07-22; First posted 2010-07-28 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Bacteremia
Keywords: pharmacokinetics
MeSH Terms: conditions — Bacteremia | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Daptomycin — once daily over 5 days

SUMMARY:
The purpose is to investigate daptomycin pharmacokinetics in critically ill patients with suspected or verified bacteremia with Gram-positive cocci undergoing combined continuous hemodiafiltration at a filtration rate of 35ml/kg/h and to establish a dose recommendation for continuous hemodiafiltration at a filtrate rate of 35ml/kg/h.

ELIGIBILITY:
Inclusion Criteria:

* male or female of 18 years or older
* females: negative pregnancy test
* Hospitalisation in the medical ICU
* High suspicion or evidence of Gram-positive infections requiring antibiotic therapy
* Subjects receiving standard antibiotic treatment for Gram-positive infection
* Evidence of renal failure
* Clinical necessity for continuous renal replacement therapy
* Written informed consent signed by the patient or a next of kin and an independent physician in case the patient is not able to sign.

Exclusion Criteria:

* Skeletal muscle disorders or CPK levels of > 2 x ULN
* History of hypersensitivity to the drug
* Participation in another study
* Subjects with a history of muscle disease
* Patients with severe liver function impairment (Child C)
* Life expectancy of less than 5 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Determination of daptomycin plasmaconcentrations and pharmacokinetics in 15 patients with gram positive infection undergoing CRRT do determine adequate dosing. | PK on days 1, 3, and 5
  15 patients are devided in 3 cohorts of 5 patients each. PK data(measured on day 1, 3 and 5) of the first 5 patients receiving daptomycin 6mg/kg/day during 5 consecutive days additionally to standard antibiotic treatment are compared with PK data of daptomycin 6mg/kg/day in healthy volunteers and dose is adapted in the next 5 patients based on these results. The same is done for the last 5 patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Intensive Care Unit, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland